CLINICAL TRIAL: NCT01340638
Title: EFFECTIVENESS OF SEAL PRESSURE IN AIRWAY OF THE CLASSIC LARYNGEAL MASK AND THE COOKGAS LARYNGEAL MASK IN ADULT PATIENTS UNDERGOING SURGERY IN AMBULATORY SETTINGS
Brief Title: Seal Pressure With Classical Laryngeal Mask and Cookgas Mask in Adult Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de Antioquia (Other)
Collaborators: Grupo de via aerea dificil universidad de antioquia (Unknown)
Responsible Party: IVAN DARIO ARENAS CORREA, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: UAntioquia SEAL- 001
Record Dates: First submitted 2011-04-19; First posted 2011-04-22 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-04

CONDITIONS: Seal Pressure
Keywords: Seal pressure; Cookgas; AirQ; LMA; supraglottic device

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cookgas (Active Comparator): This group will be assigned to use cookgas mask
  Interventions: Device: cookgas mask
- LMA mask (Active Comparator): This group will be assigned to use LMA mask
  Interventions: Device: LMA mask

INTERVENTIONS:
Device: cookgas mask — This group will be assigned to use cookgas mask
  Arms: Cookgas
Device: LMA mask — LMA mask
  Arms: LMA mask

SUMMARY:
The working hypothesis in this study is that the supraglottic device COOKGAS provides seal pressure as well or better than LMAc ™ when adult patients undergoing outpatient surgery, are sommeted to both interventions.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Patient ASA I, II and III
* Complete fast
* Ambulatory Surgery
* Time less than two hours surgically
* Supine Surgery
* Acceptance of informed consent

Exclusion Criteria:

* No acceptance of informed consent
* Pregnancy or breastfeeding
* Hemostatic alterations
* Abdominal surgery
* History of gastrointestinal reflux
* BMI over 35
* Mouth opening less than 1.5 cm
* Airway abnormalities
* Surgery in respiratory tract

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2011-06; Primary Completion 2011-11 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Seal pressures | six months
  The primary objective is to determine the effectiveness of the seal pressure between the mask COOKGAS ™ and LMAc in patients undergoing outpatient surgeries in ambulatory-based IPS, University of Antioquia (institution services health clinic) located in the city of Medellin.

CONTACTS AND LOCATIONS:
Overall Officials: IVAN D ARENAS, ANESTHETIST, Principal Investigator — Universidad de Antioquia
Locations (1):
- Ips Universitaria, Medellín, Antioquia, Colombia